CLINICAL TRIAL: NCT03686930
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation Study to Evaluate the Safety/Tolerability and Pharmacokinetics of FP-045 Administered Orally to Normal, Healthy Volunteers
Brief Title: Multiple-Dose, Dose-Escalation Study to Evaluate the Safety/Tolerability and Pharmacokinetics of FP-045
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Foresee Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: FP045C-17-001
Record Dates: First submitted 2018-04-10; First posted 2018-09-27 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Multiple Dose, Dose Escalation study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double-blind, placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 - FP-045 oral solution (Active Comparator): FP-045 powder for oral solution, will be reconstituted once daily (QD) dose, administered for 7 consecutive days.
  Interventions: Drug: Cohort 1 - FP-045 oral solution
- Cohort 1 - Placebo for FP-045 oral solution (Placebo Comparator): Placebo oral solution that is identical to the test product, but without FP-045.
  Interventions: Drug: Placebo (for FP-045 oral solution)
- Cohort 2 - FP-045 oral solution (Active Comparator): FP-045 powder for oral solution (escalated dose), will be reconstituted once daily (QD) dose, administered for 7 consecutive days.
  Interventions: Drug: Cohort 2 - FP-045 oral solution
- Cohort 2 - Placebo for FP-045 oral solution (Placebo Comparator): Placebo oral solution that is identical to the test product, but without FP-045.
  Interventions: Drug: Placebo (for FP-045 oral solution)
- Cohort 3 - FP-045 oral solution (Active Comparator): FP-045 powder for oral solution (escalated dose), will be reconstituted once daily (QD) dose, administered for 7 consecutive days.
  Interventions: Drug: Cohort 3 - FP-045 oral solution
- Cohort 3 - Placebo for FP-045 oral solution (Placebo Comparator): Placebo oral solution that is identical to the test product, but without FP-045.
  Interventions: Drug: Placebo (for FP-045 oral solution)

INTERVENTIONS:
Drug: Cohort 1 - FP-045 oral solution — FP-045 given orally with dose escalation between cohorts, based on emerging safety and pharmacokinetic (PK) data. Cohorts 2 and 3 doses to be based on the safety, tolerability, and PK data generated in the study. The dosing duration for cohorts 1-3 will be 7 consecutive days.
  Arms: Cohort 1 - FP-045 oral solution
Drug: Cohort 2 - FP-045 oral solution — FP-045 given orally with dose escalation between cohorts, based on emerging safety and pharmacokinetic (PK) data. Cohorts 2 and 3 doses to be based on the safety, tolerability, and PK data generated in the study. The dosing duration for cohorts 1-3 will be 7 consecutive days.
  Arms: Cohort 2 - FP-045 oral solution
Drug: Cohort 3 - FP-045 oral solution — FP-045 given orally with dose escalation between cohorts, based on emerging safety and pharmacokinetic (PK) data. Cohorts 2 and 3 doses to be based on the safety, tolerability, and PK data generated in the study. The dosing duration for cohorts 1-3 will be 7 consecutive days.
  Arms: Cohort 3 - FP-045 oral solution
Drug: Placebo (for FP-045 oral solution) — Participants (cohorts 1-3) will receive FP-045 oral solution matching placebo.
  Arms: Cohort 1 - Placebo for FP-045 oral solution; Cohort 2 - Placebo for FP-045 oral solution; Cohort 3 - Placebo for FP-045 oral solution

SUMMARY:
Phase I, single-center, randomized, double-blind, placebo-controlled, multiple ascending dose (MAD), study to evaluate the safety/tolerability and pharmacokinetics (PK) of FP-045 administered to normal health volunteers (NHVs). 3 cohorts of NHVs will be enrolled. Subjects in each cohort will be randomized to orally receive either FP-045 (6 subjects) or placebo (2 subjects). Subjects will receive 7 daily doses of study drug.

Subjects will be screened for study eligibility within 21 days before Day 1 and will have been admitted to the CRU on Day -1 to confirm eligibility and to undergo baseline assessments. Subjects will remain in the CRU for observation until completion of all assessments on Day 10. Subjects will return to the CRU on Day 11 for an additional PK sample, and again for an end of study (EOS) Visit on Day 14 (±2 days) for safety evaluations and collection of PK samples.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female NHV, age 18 to 55 years, inclusive (at the time of informed consent).
2. Females must be either postmenopausal for ≥1 year (or with FSH ≥ 40 mIU/mL if postmenopausal for < 1 year) or surgically sterile (having undergone bilateral tubal ligation, hysterectomy, or bilateral oophorectomy) for at least 6 months.
3. Males with female partners of childbearing potential must agree to use barrier contraceptive (i.e., condom) and their female partners must use a highly effective method of contraception from Screening through 90 days after the last dose of study drug. Males must also refrain from sperm donations during this time period.

   Males who are abstinent will not be required to use a contraceptive method unless they become sexually active.
4. The subject is, in the opinion of the Investigator, generally healthy based on assessment of medical history, physical examination, vital signs, electrocardiogram (ECG), and the results of the hematology, clinical chemistry, urinalysis, serology, and other laboratory tests.
5. Baseline laboratory test values within reference ranges based on the blood and urine samples taken at Screening and on Day -1 (before administration of the initial study drug). Out of normal ranges values may be accepted by the Investigator, if not clinically significant.
6. Nonsmoker and/or ex-smoker who has discontinued smoking and/or use of nicotine containing products for at least 6 months prior to the first dose of study drug
7. Body mass index between 18 and 30 kg/m2, inclusive
8. Written informed consent obtained Ability to communicate well with the Investigator, in the local language, and to understand and comply with the requirements of the study.

Exclusion Criteria:

1. History or presence of any clinically significant neurological, metabolic, gastrointestinal, endocrinological (in particular diabetes or pre-diabetes), cardiovascular, hematological, hepatic, immunological, renal, respiratory, chronic infections, psychiatric, or genitourinary abnormalities or diseases. Note: NHVs with a history of uncomplicated kidney stones or asthma may be enrolled in the study at the discretion of the Investigator.
2. History of malignant neoplastic disease, with the following exceptions:

   1. Adequately treated non-melanomatous skin carcinoma
   2. Female with a history of benign cervical carcinoma neoplasia if compliant with surveillance and treatment as recommended by her physician
3. Mentally or legally incapacitated, has significant emotional problems at Screening or expected during the conduct of the study, or has a history of a clinically significant psychiatric disorder within the last 5 years. Note: NHVs who have had situational depression may be enrolled in the study at the discretion of the Investigator.
4. The subject has a history of severe drug allergy or hypersensitivity or food allergy, including anaphylaxis.
5. The subject has had surgery or trauma with significant blood loss within the last 3 months prior to the first dose of study drug.
6. The subject has donated blood more than 1 unit (500 mL) with 4 weeks prior to the first dose of study drug.
7. Fever (body temperature >38°C) or symptomatic viral or bacterial infection within 2 weeks prior to Screening
8. Blood pressure >140/90 mm Hg or heart rate >100 beats per minute at Screening or at Day -1. Vitals may be repeated up to 2 times for the purpose of eligibility.
9. Clinically significant laboratory abnormalities including:

   1. Impaired renal function (serum creatinine levels >ULN) at Screening; estimated creatinine clearance (CrCl) of <80 mL/min
   2. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) laboratory values >1.2 × upper normal limits
10. Clinically significant abnormality on ECG performed at Screening or prior to administration of the initial dose of study drug. (Screening ECG conduction intervals must be 10. Clinically significant abnormality on ECG performed at Screening or prior to administration of the initial dose of study drug. (Screening ECG conduction intervals must be within gender specific normal ranges [QT interval corrected for heart rate [QTc] males ≤450 msec and females ≤470 msec].)
11. Positive test for hepatitis C antibody, hepatitis B surface antigen, or human immunodeficiency virus antibody at Screening
12. Positive screen for drugs with a high potential for abuse (amphetamine, cannabinoid, cocaine, morphine, and phencyclidine) at Screening and Study Day -1.
13. Consumed food or drink containing grapefruit juice within 72 hours before start of dosing or expected to do so through EOS/ET
14. Consumed alcohol within 72 hours before start of dosing through EOS/ET.
15. Received any previous FP-045 or has taken any investigational product within 30 days or 5 half-lives (whichever is longer) prior to the first dose of study drug.
16. Female who is breastfeeding or has a positive pregnancy test
17. Unwilling or unable to comply with the requirements of this protocol, including the presence of any condition (physical, mental, or social) that is likely to affect the subject's return for the scheduled EOS Visit
18. The subject has taken prescription medications within 2 weeks (or within 5 half-lives, whichever is longer) or nonprescription medication, herbal remedies, vitamins or minerals within 1 week prior to the administration of the initial dose of study drug and continuing throughout the study until the final study visit. Note: There may be certain medications that are permitted at the discretion of the Investigator and Sponsor (including paracetamol/ acetaminophen, which may be used for minor ailments during the course of the study without prior consultation with the Sponsor's Medical Monitor).
19. The subject exercises extensively (e.g. marathon, triathlon or other similar high energetic sports). In general, subjects should refrain from sporting for at least 4 days before participation in the study until the EOS/ET visit.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2018-05-27 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Change in baseline measures for vital sign parameters [safety/tolerability] | 14 days ± 2 days
  Outcome Measures units of measure include weight in kilograms.
Change in baseline measures for ECG parameters [safety/tolerability] | 14 days ± 2 days
  T wave
Change in baseline measures for clinical laboratory test [safety/tolerability] | 14 days ± 2 days
  Number of Participants with Abnormal Laboratory Values. Blood will be drawn to measure the chemistry of the blood prior to and after dosing.
Number of participants with treatment-emergent ECG abnormalities [safety/tolerability]. | 14 days ± 2 days
Number of participants with treatment-emergent AEs [safety/tolerability]. | 14 days ± 2 days
Number of participants with treatment-emergent AEs leading to premature discontinuation of study drug [safety/tolerability]. | 14 days ± 2 days
Number of participants with treatment-emergent SAEs [safety/tolerability]. | 14 days ± 2 days
Change in baseline measures for vital sign parameters [safety/tolerability] | 14 days ± 2 days
  Outcome Measures units of measure include height in meters.
Change in baseline measures for vital sign parameters [safety/tolerability] | 14 days ± 2 days
  Outcome Measures units of measure include blood pressure both systolic and diastolic will be measured.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile (Cmax) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
  Cmax (maximum plasma concentration) -first and last doses (Day 1 and Day 7) of FP-045 will be measured.
Pharmacokinetic (PK) profile (Tmax) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
  Tmax (time to maximum plasma concentration) -first and last doses (Day 1 and Day 7) of FP-045 will be measured.
Pharmacokinetic (PK) profile (AUC0-24) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
  AUC0-24 (area under the curve from time 0 to 24 hours postdose) - first dose (Day 1) of FP-045 will be measured.
Pharmacokinetic (PK) profile (Cavg) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
  Cavg (average plasma concentration over the dosing interval) = AUC0-24/τ, where τ is the dosing interval - last dose (Day 7) of FP-045 will be measured.
Pharmacokinetic (PK) profile (accumulation ratio of AUC0-24) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
  Accumulation ratio of AUC0-24 (Day 7)/AUC0-24 (Day 1) of FP-045 will be measured.
Pharmacokinetic (PK) profile (AUC[0-24]) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
  AUC[0-24](area under the curve over the dosing interval) - Day 7 of FP-045 will be measured.
Other pharmacokinetic (PK) profiles measured include t1/2 (terminal half-life) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
Other pharmacokinetic (PK) profiles measured include CL/F (apparent clearance) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
Other pharmacokinetic (PK) profiles measured include Vz/F (apparent volume of distribution) following multiple, escalating oral doses of FP-045. | 14 days ± 2 days
Other pharmacokinetic (PK) profiles measured include elimination rate constant following multiple, escalating oral doses of FP-045. | 14 days ± 2 days

CONTACTS AND LOCATIONS:
Overall Officials: David Lau, Ph.D., Study Director — Foresee Pharma
Locations (1):
- Nucleus Networks, Melbourne, Australia

IPD SHARING:
Plan to Share IPD: Undecided